CLINICAL TRIAL: NCT00854581
Title: Prospective Study of the Molecular Characteristics of Sensitive and Resistant Disease in Patients With HTLV-I Associated Adult T Cell Leukemia Treated With Zidovudine (AZT) Plus Interferon Alpha-2b
Brief Title: Zidovudine, Interferon Alfa-2b, PEG-Interferon Alfa-2b in Patients With HTLV-I Associated Adult T-Cell Leukemia/Lymphoma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator Decision
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Juan C. Ramos, Associate Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20070805; SCCC-2007055 (Other: UM/Sylvester Comprehensive Cancer Center); 5P01CA128115-02 (NIH)
Record Dates: First submitted 2009-02-28; First posted 2009-03-03 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2017-12

CONDITIONS: Lymphoma; Precancerous/Nonmalignant Condition
Keywords: recurrent adult T-cell leukemia/lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; HTLV-1 infection
MeSH Terms: conditions — Lymphoma; Precancerous Conditions; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; HTLV-I Infections | interventions — peginterferon alfa-2b; Interferon alpha-2; Valproic Acid; Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Induction (Up to Day 21) (Experimental): For one cycle, up to Day 21. All participants are enrolled to induction therapy phase, then move to the maintenance therapy phase if they achieve complete response (PR) or partial response (PR). Participants who achieve a clinical CR at Day 14 response assessment will go on to Part 1 maintenance therapy. Patients who achieve a PR will receive 7 more days of induction therapy and then go on to Part 1 Maintenance Therapy.:
  * Zidovudine:
    * Days 1-2: 1.5 grams intravenously (IV) twice daily
    * Days 3-21: 1.5 grams IV twice daily
  * Interferon alfa-2b (IFN):
    * 5 10 million units (mu) intravenously twice daily
  Interventions: Biological: Interferon alfa-2b; Drug: Zidovudine
- Part 1 Maintenance (Up to Day 60) (Experimental): From Treatment Day 14 or 21 to start of Month 3 (Day 60). Study participants move on to Part 1 Maintenance Therapy only if they achieve complete response (CR) or partial response (PR) after induction therapy. Restaging and molecular evaluation of disease at start of Month 3:
  * Zidovudine: 600 mg orally twice daily in all phases of Maintenance Therapy
  * PEG-Interferon alfa-2b: 1.5 ug/kg subcutaneously (SQ) once weekly
  * Participants then proceed to Part 2 maintenance.
  Interventions: Biological: PEG-interferon alfa-2b; Drug: Zidovudine
- Part 2A Maintenance (Up to 12 Months) (Experimental): Participants achieving a CR with undetectable clonal disease. Participants will receive therapy for as long as response is maintained:
  * Zidovudine: 600 mg orally twice daily
  * PEG-Interferon alfa-2b: 1.5 ug/kg subcutaneously (SQ) once weekly
  Interventions: Biological: PEG-interferon alfa-2b; Drug: Zidovudine
- Part 2B Maintenance (Up to 12 Months) (Experimental): Participants achieving a CR with minimal residual disease (by multiplex PCR) or PR in Part 1:
  * Zidovudine: 600 mg or 300 mg orally twice daily, per protocol
  * PEG-Interferon alfa-2b: 1.5 ug/kg subcutaneously (SQ) once weekly, per protocol
  * Valproic acid, 250 mg orally twice daily, per protocol
  Interventions: Biological: PEG-interferon alfa-2b; Drug: Valproic Acid; Drug: Zidovudine

INTERVENTIONS:
Biological: PEG-interferon alfa-2b — Administered subcutaneously.
  Other Names: PEG-IFN-alfa2b
  Arms: Part 1 Maintenance (Up to Day 60); Part 2A Maintenance (Up to 12 Months); Part 2B Maintenance (Up to 12 Months)
Biological: Interferon alfa-2b — Administered intravenously.
  Arms: Induction (Up to Day 21)
Drug: Valproic Acid — Administered orally.
  Other Names: Depakene
  Arms: Part 2B Maintenance (Up to 12 Months)
Drug: Zidovudine — Administered intravenously during Induction Therapy; orally during Maintenance Therapy in all Phases (1, 2A and 2B).
  Other Names: Retrovir; AZT

SUMMARY:
RATIONALE: Human T-cell lymphotropic virus type 1 (HTLV-1) can cause cancer. Zidovudine is an antiviral drug that acts against the human T-cell lymphotropic virus type 1. Giving zidovudine, interferon alfa-2b, and PEG-interferon alfa-2b together may stimulate the immune system and slow down or keep the cancer cell from growing.

PURPOSE: This clinical trial is studying how well giving zidovudine together with interferon alfa-2b and PEG-interferon alfa-2b works in treating patients with human T-cell lymphotropic virus type 1-associated adult T-cell leukemia/lymphoma.

DETAILED DESCRIPTION:
OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive zidovudine IV twice daily on days 1-14, and recombinant interferon alfa-2b IV twice daily on days 3-14. Patients achieving clinical complete response (CR) proceed to part 1 maintenance therapy; patients achieving partial response (PR) receive another 7 days of zidovudine and recombinant interferon alfa-2b and then proceed to part 1 maintenance therapy.
* Part 1 maintenance therapy: Patients receive oral zidovudine twice daily and PEG-interferon alfa-2b subcutaneously (SC) once weekly, beginning on day 14 or 21 and continue to day 60. Patients are evaluated after completion of part 1 maintenance therapy and proceed to part 2 maintenance therapy.
* Part 2 maintenance therapy: Patients achieving CR with undetectable clonal disease proceed to group A; patients achieving CR with minimal residual disease (by PCR) or PR proceed to group B.

  * Group A: Patients receive oral zidovudine twice daily and PEG-interferon alfa-2b SC once weekly. Treatment continues in the absence of disease progression or unacceptable toxicity.
  * Group B: Patients receive oral zidovudine twice daily and PEG-interferon alfa-2b SC once weekly for 12 weeks and undergo reevaluation. Patients in continued CR with minimal residual disease or stable PR receive oral valproic acid twice daily, PEG-interferon alfa-2b SC once weekly, and oral zidovudine twice daily for 6 months. At that point (month 9) patients with no detectable clonal disease continue their previous treatment, while patients with minimal residual disease receive PEG-interferon alfa-2b SC and oral zidovudine twice daily in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline, days 1 and 2, and months 3, 6, and 12 for protein, genomic DNA, and RNA analysis. Baseline molecular characteristics of the tumor and tumor response to treatment is assessed.

After completion of study treatment, patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria

* Any stage, histologically or cytological documented adult T-cell leukemia/lymphoma (ATLL), leukemic types only (smoldering, chronic or acute). See Appendix I for definitions of the clinical subtypes.
* Patients who have received prior treatment, including zidovudine and/or IFN, are eligible, provided that zidovudine/IFN therapy did not result in progressive disease.
* Documented HTLV-I infection: documentation may be serologic assay (ELISA, Western blot) and confirmed to be HTLV-I rather than HTLV-2 by differential Western blot (e.g., Genelabs Diagnostics HTLV Blot 2.4) or PCR.
* Measurable or evaluable disease.
* Age 18 or older.
* Karnofsky performance status ≥ 50%.
* Patients must have adequate end organ and bone marrow function as defined below:

  * Absolute neutrophil count ≥ 1,000 cells/mm3 and platelets ≥ 50,000 cells/mm3 unless cytopenias are secondary to ATLL.
  * Adequate hepatic function: (transaminase ≤ 7 times the upper limit of normal, total bilirubin < 2.0), unless secondary to hepatic infiltration with lymphoma. If the elevated bilirubin is felt to be secondary to Indinavir or Atazavinir therapy (anti-HIV medications), patients will be allowed to enroll on protocol if the total bilirubin is ≤ 3.5 mg/dl provided that the direct bilirubin is normal.
  * Creatinine < 2.0 unless due to lymphomatous infiltration.
* Patients who are HIV+ are also eligible.
* Females with childbearing potential must have a negative serum pregnancy test within 72 hours of entering into the study. Males and females must agree to use adequate birth control if conception is possible during the study. Women must avoid pregnancy and men avoid fathering children while in the study.
* Able to give consent.
* Patients already receiving erythropoietin or granulocyte-colony stimulating factor (G-CSF) are eligible.

Exclusion Criteria

* Concurrent active malignancies, with the exception of in situ carcinoma of the cervix, non-metastatic, non-melanomatous skin cancer, or Kaposi's sarcoma not requiring systemic chemotherapy.
* Grade 3 or 4 cardiac failure and/or ejection fraction < 50%.
* Psychological, familial, sociological or geographical conditions that do not permit treatment and/or medical follow-up required to comply with the study protocol.
* Patients may not be receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast-feeding women.
* Hypersensitivity to interferon alpha-2b, peginterferon alpha-2b, zidovudine or any component of the formulation
* Autoimmune or viral hepatitis or decompensated liver disease unless due to lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-11; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Ramos, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction + Maintenance: All participants are enrolled to induction therapy first, then move to the maintenance therapy Parts 1 and 2A or 2B if they achieve complete response (PR) or partial response (PR).
Period: Induction (Up to Day 21)
Arm/Group | Induction + Maintenance
Started | 13
Completed | 7
Not Completed | 6
Not completed — Lack of Efficacy | 4
Not completed — Death | 1
Not completed — Physician Decision | 1
Period: Part 1 Maintenance (Up to Day 60)
Arm/Group | Induction + Maintenance
Started | 7
Completed | 5
Not Completed | 2
Period: Part 2 Maintenance (Up to 12 Months)
Arm/Group | Induction + Maintenance
Started | 5
Completed | 2
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Induction + Maintenance
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 0
  More than one race | 2
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Brazil | 1
  Dominican Republic | 1
  Haiti | 3
  Jamaica | 5
  St. Croix | 1
  Trinidad | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Clinical Response to Protocol Therapy Who Lack IRF-4 and/or c-Rel Expression.
Description: Number of patients achieving clinical response (complete response (CR) + partial response (PR)) who lack interferon regulatory factor 4 (IRF-4) or c-Rel biomarker expression. Treatment response was assessed according to the International Consensus Review's adult T-cell leukemia/lymphoma (ATLL) consensus report by Tsukasaki et al published in the Journal of Clinical Oncology (JCO) in 2009.
  For imaging, Cheson criteria was used to assess response:
  * Complete response (CR): Disappearance of all clinical, microscopic, and radiographic evidence of disease. All lymph nodes regressed to normal size (≤ 1.5 cm), and previously involved nodes that were 1.1 to 1.5 cm decreased to ≤ 1.0 cm. In addition, abnormally elevated peripheral blood absolute lymphocyte count (ALC) < 4 x 10^9 /L.
  * Partial response (PR): ≥ 50% reduction in measurable disease and abnormal lymphocyte count in peripheral blood.
  * CR or PR had to persist for a period of at least 4 weeks.
Time Frame: Up to 12 months post-initiation of protocol therapy
Population: All participants who had a treatment response (PR or CR)
Measure: Number; unit: participants
Arm/Group | Induction + Maintenance
Number analyzed (Participants) | 6
participants
  Participants with tumors lacking IRF-4 | 5
  Participants with tumors lacking c-Rel: number analyzed (Participants) | 4
  Participants with tumors lacking c-Rel | 2

2. Primary Outcome: Presence of Minimal Residual Disease at 3 and 6 Months of Maintained Remission and at 1 Year Post Initiation of Therapy
Description: Number of participants achieving complete response (CR) with minimal residual disease at 3, 6 and 12 months post-initiation of protocol therapy. Treatment response was assessed according to the International Consensus Review's adult T-cell leukemia/lymphoma (ATLL) consensus report by Tsukasaki et al published in the Journal of Clinical Oncology (JCO) in 2009.
  For imaging, Cheson criteria was used to assess response:
  * Complete response (CR): Disappearance of all clinical, microscopic, and radiographic evidence of disease. All lymph nodes regressed to normal size (≤ 1.5 cm), and previously involved nodes that were 1.1 to 1.5 cm decreased to ≤ 1.0 cm. In addition, abnormally elevated peripheral blood absolute lymphocyte count (ALC) < 4 x 10^9 /L.
  * Partial response (PR): ≥ 50% reduction in measurable disease and abnormal lymphocyte count in peripheral blood.
  * CR or PR had to persist for a period of at least 4 weeks.
Time Frame: 3, 6 and 12 months.
Population: Participants who achieved CR with minimal residual disease in Part 1 Maintenance therapy at Month 3 and moved on the Part 2B maintenance for up to 12 months.
Measure: Number; unit: participants
Groups:
- Part 2B Maintenance (Up to 12 Months): Participants achieving a CR with minimal residual disease (by multiplex PCR) or PR in Part 1:
  * Zidovudine: 600 mg or 300 mg orally twice daily, per protocol
  * PEG-Interferon alfa-2b: 1.5 ug/kg subcutaneously (SQ) once weekly, per protocol
  * Valproic acid, 250 mg orally twice daily, per protocol
  Valproic Acid: Administered orally.
Arm/Group | Part 2B Maintenance (Up to 12 Months)
Number analyzed (Participants) | 3
participants
  3 months, CR w/minimal residual disease | 3
  6 months, CR w/minimal residual disease | 1
  12 months, CR w/minimal residual disease | 0

3. Primary Outcome: Expressions of c-Rel, IRF-4 and Other Molecular Events in Participants
Description: Expressions of c-Rel, IRF-4 or other molecular events (p53, p16 mutations) including expansion of novel clones obtained at time of relapse will be compared to baseline data using paired t-test.
Time Frame: At time of relapse or disease progression, assessed up to 12 months
Population: Study participants were tested for these markers at baseline, but only IRF4 was re-tested at relapse
Measure: Number; unit: participants
Arm/Group | Induction + Maintenance
Number analyzed (Participants) | 12
participants
  Baseline IRF-4 Expression, Positive | 3
  Baseline IRF-4 Expression, Negative | 9
  IRF-4 Expression at Relapse, Newly Positive: number analyzed (Participants) | 4
  IRF-4 Expression at Relapse, Newly Positive | 2
  Baseline c-Rel Expression, Faintly Positive: number analyzed (Participants) | 8
  Baseline c-Rel Expression, Faintly Positive | 3
  Baseline c-Rel Expression, Positive: number analyzed (Participants) | 8
  Baseline c-Rel Expression, Positive | 2
  Baseline c-Rel Expression, Negative: number analyzed (Participants) | 8
  Baseline c-Rel Expression, Negative | 3
  Baseline p53 Expression, Positive: number analyzed (Participants) | 6
  Baseline p53 Expression, Positive | 1
  Baseline p53 Expression, Negative: number analyzed (Participants) | 6
  Baseline p53 Expression, Negative | 5
  Baseline p15/16 alterations, homozygous deletion: number analyzed (Participants) | 5
  Baseline p15/16 alterations, homozygous deletion | 1
  Baseline p15/16 alterations, heterozygous deletion: number analyzed (Participants) | 5
  Baseline p15/16 alterations, heterozygous deletion | 2
  Baseline p15/16 alterations, no deletions: number analyzed (Participants) | 5
  Baseline p15/16 alterations, no deletions | 2

4. Primary Outcome: Number of Participants Exhibiting NF-kB Inhibition Upon Treatment With AZT in Vivo
Description: Number of patients exhibiting NF-kb inhibition upon treatment with AZT in vivo. Investigation of whether AZT functions as an inhibitor of nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kB) in vivo by analyzing serially collected leukemic samples during the first 48 hours of treatment with AZT only. The investigators will report the number of participants exhibiting NF-kB inhibition upon treatment with AZT in vivo and correlate with response using two-sample t-test.
Time Frame: During 48 hours of first AZT therapy
Population: Participants receiving Zidovudine (AZT) therapy who achieved complete response (CR) or partial response (PR).
Measure: Number; unit: participants
Groups:
- Induction (Up to Day 21): For one cycle, up to Day 21. All participants are enrolled to induction therapy phase, then move to the maintenance therapy phase if they achieve complete response (PR) or partial response (PR). Participants who achieve a clinical CR at Day 14 response assessment will go on to Part 1 maintenance therapy. Patients who achieve a PR will receive 7 more days of induction therapy and then go on to Part 1 Maintenance Therapy.:
  * Zidovudine:
    * Days 1-2: 1.5 grams intravenously (IV) twice daily
    * Days 3-21: 1.5 grams IV twice daily
  * Interferon alfa-2b (IFN):
    * 5 10 million units (mu) intravenously twice daily
  Interferon alfa-2b: Administered intravenously.
  Zidovudine: Administered intravenously during Induction Therapy; orally during Maintenance Therapy in all Phases (1, 2A and 2B).
Arm/Group | Induction (Up to Day 21)
Number analyzed (Participants) | 4
participants
  CR with Decrease in NF-kB Complex (p50 complexes) | 1
  CR with no clear effect NF-kB | 1
  PR with Decrease in p50, and Increase in p65 | 1

5. Primary Outcome: The Effect of Valproic Acid Therapy on Persistence of Clonal Disease in Patients Who Achieve Clinical Remission
Description: Number of participants achieving a molecular remission after starting valproic acid as evidenced by disappearance of T-cell clonality as measured by gene rearrangement studies using multiplex PCR
Time Frame: 3, 6 and 12 months.
Population: Participants achieving CR or PR in Part 1 Maintenance and moving on to Part 2B Maintenance therapy
Measure: Number; unit: participants
Arm/Group | Part 2B Maintenance (Up to 12 Months)
Number analyzed (Participants) | 3
participants
  3 months, CR or PR, with molecular remission | 0
  6 months, CR with molecular remission | 1
  9 months, CR with molecular remission | 1
  12 months, CR with molecular remission | 1

6. Secondary Outcome: Failure-free Survival (FFS)
Description: Failure-free survival is the elapsed time from the date of initiation of study treatment until date of documented disease progression, relapse after response, or death from any cause. For patients alive and free of relapse or progression, follow-up time was censored at the last documented date of failure-free status.
Time Frame: From date of treatment initiation until date of documented disease progression, relapse after response, or death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction + Maintenance
Number analyzed (Participants) | 13
months | 2.7 [1.0 to 6.9]

7. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is the elapsed time from the date of initiation of study treatment until date of death from any cause. In the absence of death, the follow-up was censored at date of last contact.
Time Frame: From date of treatment initiation until date of death, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction + Maintenance
Number analyzed (Participants) | 13
months | 7.8 [2.5 to 46.6]

ADVERSE EVENTS:
Groups:
- Induction Therapy: For one cycle, up to Day 21. All participants are enrolled to induction therapy phase, then move to the maintenance therapy phase if they achieve complete response (PR) or partial response (PR). Participants who achieve a clinical CR at Day 14 response assessment will go on to Part 1 maintenance therapy. Patients who achieve a PR will receive 7 more days of induction therapy and then go on to Part 1 Maintenance Therapy.:
  * Zidovudine:
    * Days 1-2: 1.5 grams intravenously (IV) twice daily
    * Days 3-21: 1.5 grams IV twice daily
  * Interferon alfa-2b (IFN):
    * 5 10 million units (mu) intravenously twice daily
- Part 1 Maintenance: From Treatment Day 14 or 21 to start of Month 3 (Day 60). Study participants move on to Part 1 Maintenance Therapy only if they achieve complete response (CR) or partial response (PR) after induction therapy. Restaging and molecular evaluation of disease at start of Month 3:
  * Zidovudine: 600 mg orally twice daily in all phases of Maintenance Therapy
  * PEG-Interferon alfa-2b: 1.5 ug/kg subcutaneously (SQ) once weekly
  * Participants then proceed to Part 2 maintenance.
- Part 2A Maintenance: Participants achieving a CR with undetectable clonal disease. Participants will receive therapy for as long as response is maintained:
  * Zidovudine: 600 mg orally twice daily
  * PEG-Interferon alfa-2b: 1.5 ug/kg subcutaneously (SQ) once weekly
- Part 2B Maintenance: Participants achieving a CR with minimal residual disease (by multiplex PCR) or PR in Part 1:
  * Zidovudine: 600 mg or 300 mg orally twice daily, per protocol
  * PEG-Interferon alfa-2b: 1.5 ug/kg subcutaneously (SQ) once weekly, per protocol
  * Valproic acid, 250 mg orally twice daily, per protocol
Arm/Group | Induction Therapy | Part 1 Maintenance | Part 2A Maintenance | Part 2B Maintenance
All-Cause Mortality (participants affected / at risk) | 5/13 | 2/7 | 0/2 | 1/3
Serious Adverse Events (participants affected / at risk) | 2/13 | 1/7 | 1/2 | 1/3
Other Adverse Events (participants affected / at risk) | 12/13 | 2/7 | 1/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Therapy (N=13) | Part 1 Maintenance (N=7) | Part 2A Maintenance (N=2) | Part 2B Maintenance (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection - Other (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infection, Catheter-related (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Therapy (N=13) | Part 1 Maintenance (N=7) | Part 2A Maintenance (N=2) | Part 2B Maintenance (N=3)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Edema: Head and Neck (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 3 (7) | 1 (1) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection, Bladder (urinary) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection, normal ANC, Catheter-related (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection, Urinary tract NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 1 (1) | 1 (1)
Lymphatics - Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (7) | 0 (0) | 1 (2) | 2 (2)
Neutrophils (Blood and lymphatic system disorders) | 4 (6) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scleral necrosis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes